CLINICAL TRIAL: NCT04474964
Title: Focal Radiotherapy Plus Low Dose Craniospinal Irradiation Followed by Adjuvant Chemotherapy in WNT Subgroup Medulloblastoma.
Brief Title: Focal Radiotherapy Plus Low Dose Craniospinal Irradiation Followed by Adjuvant Chemotherapy in WNT Medulloblastoma.
Acronym: FOR-WNT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3468
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Medulloblastoma, WNT-activated
Keywords: WNT medulloblastoma; low dose craniospinal irradiation; overall survival; long term toxicities
MeSH Terms: conditions — Medulloblastoma | interventions — Craniospinal Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Dose Craniospinal Irradiation (Experimental): WNT subgroup medulloblastoma patients accrued in the study will be treated with Low-dose Craniospinal Irradiation (18Gy/10fx) plus focal conformal tumor-bed boost (36Gy/20fx) for total primary-site dose of 54Gy/30fx over 6-weeks. Followed by adjuvant multi-agent systemic chemotherapy which will be initiated 4-6 weeks after completion of radiotherapy provided the ANC >1500 and platelet count >1,00,000. A total of 6 cycles of alternating chemotherapy every 4-weekly will be planned as per our standard practice using CET protocol.
  Interventions: Radiation: Low dose Craniospinal Irradiation plus Focal Radiotherapy

INTERVENTIONS:
Radiation: Low dose Craniospinal Irradiation plus Focal Radiotherapy — The intervention arm of the study is to prospectively evaluate disease-related outcomes of low-dose CSI plus focal radiotherapy without concurrent chemotherapy followed by standard 6-cycles of adjuvant systemic chemotherapy in WNT-pathway medulloblastoma.

SUMMARY:
This clinical study is going to be done on a type of brain tumor in children called Medulloblastoma. The WNT pathway type of medulloblastoma is considered to be low risk and have the best outcomes in terms of survival. With the current standard of care for this type of medulloblastoma it is believed by the investigators that we are over treating the disease and increasing the long term side effects of these children. Several groups in the world are testing de-intensification of treatment in this favourable subset of children who experience long term late side effects of therapy. By reducing the dose to the craniospinal axis and keeping the total tumor bed dose the same in this study the investigators are expecting to reduce some of the late side effects of craniospinal irradiation without compromising disease control and survival.

DETAILED DESCRIPTION:
WNT pathway medulloblastomas have the best prognosis amongst all four subgroups with 5-year overall survival exceeding 90%. Overall medulloblastoma is more common in males. They can occur at all ages, but, are uncommon in infants. They are mostly uniform in their genetic aberrations, histological pattern, and clinical presentation. The WNT pathway is involved in regulating embryonal development in the brain. They are frequently described as having CTNNB1 mutations, nuclear immunohistochemical staining for β-catenin, and monosomy six (deletion of one copy of chromosome 6 in the tumor). Thus monosomy 6 in conjunction with nuclear β-catenin accumulation is considered a sensitive and specific marker for WNT pathway medulloblastoma they are typically located in the midline vermian region filling up the fourth ventricle and infiltrating the brain stem consistent with their proposed cell of origin from the dorsal brainstem nuclei. The immediate impact of enhanced understanding of molecular biology has led to biologically driven next-generation clinical trials in newly diagnosed medulloblastoma. Given the excellent long-term survival outcomes in WNT-pathway medulloblastoma and potential for significant late toxicities with currently prevalent doses of CSI (23.4-36Gy), it has been hypothesized that further reduction of dose or in certain cases avoidance of CSI would translate into reduction in late morbidity of treatment.

In our first generation FOR-WNT study, the investigators had avoided upfront CSI and treated the tumor-bed alone with focal conformal radiotherapy in low-risk WNT-pathway medulloblastoma followed by 6-cycles of adjuvant systemic chemotherapy. However, early experience from our own study and similar results from another study (primary chemotherapy approach completely avoiding radiotherapy) suggests an unduly increased risk of relapse - spinal leptomeningeal or supratentorial if CSI is avoided and local recurrence at primary site too if radiation is completely avoided. Given the excellent long-term survival outcomes in WNT-pathway medulloblastoma treated with currently prevalent doses of CSI (23.4-36Gy), presence of significant late toxicities with such doses, but the increased risk of relapse with avoidance of CSI and/or local irradiation, the investigators hypothesize that further moderate reduction of CSI dose to 18Gy/10fx keeping the primary-site dose to 54Gy/30fx would translate into a meaningful reduction in late morbidity of treatment without compromising disease control or survival. Thus, the investigators herewith propose the second-generation study (FOR-WNT 2) to include low-dose CSI (18Gy/10fx) plus tumor-bed boost (36Gy/20fx) for a total primary site dose of 54Gy/30fx without concurrent chemotherapy followed by standard 6-cycles of adjuvant systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 3 years and less than 16 years.
* Newly diagnosed WNT pathway medulloblastoma.
* Post-surgery residual disease less than 1.5 cm2 on post-operative MRI brain.
* No evidence of metastatic disease in the brain, spine or cerebral spinal fluid (CSF) assessed by MRI of the brain/spine and lumbar puncture for CSF cytology.
* Fit for initiation of adjuvant treatment within 6-weeks of surgery

Exclusion Criteria:

* Age Less than 3 and more than 16 years.
* Molecular subgroup other than WNT pathway.
* Post-surgery residual disease more than 1.5cm2 on post-operative imaging.
* Evidence of any metastatic disease in the brain, spine or CSF.
* Previous history of radiotherapy or chemotherapy prior to study enrollment.
* Not fit for initiation of adjuvant treatment within 6 weeks of surgery.
* Not willing for consent/assent.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival will be analysed using using the product-limit method of Kaplan-Meier and compared using the log-rank test. | 5 years
  Measure Relapse-free survival in WNT medulloblastoma treated with low-dose CSI plus focal radiotherapy without concurrent chemotherapy followed by standard 6-cycles of adjuvant systemic chemotherapy. Relapse free survival will be calculated from the date of surgery till the first documented clinico-radiological evidence of relapse (recurrence/progression).
Overall Survival of Participants will be analysed using the product-limit method of Kaplan-Meier and compared using the log-rank test. | 5 years
  Measure Overall survival in WNT medulloblastoma treated with low-dose CSI plus focal radiotherapy without concurrent chemotherapy followed by standard 6-cycles of adjuvant systemic chemotherapy.Overall survival will be measured from the date of diagnosis till death from any cause.

SECONDARY OUTCOMES:
Neuro-cognitive function of Participants will be analysed longitudinally over time using linear regression model with time-test for trend | 5 years
  Neurocognitive Outcome will be assessed using Wechsler scale for children by comparing pre-radiotherapy result with assessment done 3-6 months after radiotherapy, at 1-year post-treatment, and annually thereafter till 5-years.
Growth Hormone levels of Participants will be analysed longitudinally over time using linear regression model with time-test for trend. | 5 years
  Serial Serum growth hormone(ng/ml) levels will be done by comparing pre-radiotherapy levels with biochemical assessment done 3-6 months after radiotherapy, at 1-year post-treatment and annually thereafter for 5-years.
Thyroid function levels of Participants will be analysed longitudinally over time using linear regression model with time-test for trend. | 5 years
  Serial Thyroid function levels : TSH , T3, T4 levels will be done by comparing pre-radiotherapy levels with biochemical assessment done 3-6 months after radiotherapy, at 1-year post-treatment and annually thereafter for 5-years.
Cortisol levels of Participants will be analysed longitudinally over time using linear regression model with time-test for trend. | 5 years
  Serial Cortisol levels (mcg/dl) will be done by comparing pre-radiotherapy levels with biochemical assessment done 3-6 months after radiotherapy, at 1-year post-treatment and annually thereafter for 5-years.
Sex Hormone levels of Participants will be analysed longitudinally over time using linear regression model with time-test for trend. | 5 years
  Sex Hormone levels will be done by comparing pre-radiotherapy levels with biochemical assessment done 3-6 months after radiotherapy, at 1-year post-treatment and annually thereafter for 5-years.
Pure tone Audiometry of Participants will be analysed longitudinally over time using linear regression model with time-test for trend. | 5 years
  Hearing assessment will be done by comparing baseline results with hearing assessment 3-6 months after radiotherapy, at 1-year post-treatment, and annually thereafter for 5-years.

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No